CLINICAL TRIAL: NCT01229618
Title: A Phase 1 Ascending-dose Study to Assess the Safety and Tolerability and Imaging Potential of Hyperpolarized Pyruvate (13C) Injection in Subjects With Prostate Cancer
Brief Title: Hyperpolarized Pyruvate Injection in Subjects With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Charles Ryan, Clinical Professor of Medicine and Urology, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 085517
Record Dates: First submitted 2010-10-13; First posted 2010-10-28 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 0.14 ml/kg bw - hyperpolarized pyruvate
  Interventions: Drug: Hyperpolarized Pyruvate (13C) injection
- 2 (Experimental): 0.28 ml/kg bw - hyperpolarized pyruvate
  Interventions: Drug: Hyperpolarized Pyruvate (13C) injection
- 3 (Experimental): 0.43 ml/kg bw - hyperpolarized pyruvate
  Interventions: Drug: Hyperpolarized Pyruvate (13C) injection

INTERVENTIONS:
Drug: Hyperpolarized Pyruvate (13C) injection — single hyperpolarized pyruvate IV (intravenous) injection followed by MR imaging scans (MRI and MRSI)
  Other Names: [1-13C]pyruvic acid; AH111710

SUMMARY:
Current imaging options do not assess prostate cancer well. This study will combine two magnetic resonance imaging modalities, MRI and MRSI, in order to determine the utility to physicians and patients with prostate cancer in making treatment decisions and seeing how well various types of treatment work. Hyperpolarized pyruvate (13C) is an investigational product that may enhance the imaging capability of MRI and MRSI. Hyperpolarized pyruvate will be injected into the body to determine how it is metabolized and how it's metabolism can be assessed using MR imaging.

The purpose of this study is to determine the safety and metabolism of hyperpolarized pyruvate in humans, and how this can be used to increase the effectiveness of MR imaging with regards to patient care.

DETAILED DESCRIPTION:
This is a phase 1 clinical study of an investigational medicinal product (IMP), hyperpolarized Pyruvate (13C) Injection. The study includes the acquisition of magnetic resonance (MR) data and will be performed in men with prostate cancer and intact prostates.

A standard dose-escalation design will be used; initially, 6 subjects will receive IMP at each dose level. As data on both the dynamics of arrival of the IMP and potential imaging efficacy are needed at each dose level, requiring the use of separate MR acquisition sequences, a modified 3+3 design will be applied in each dose cohort. The first 3 subjects will undergo dynamic 13C imaging to define the kinetics of delivery and metabolism of IMP, and the second 3 subjects will undergo 13C MR spectroscopic imaging (MRSI) to obtain 3-dimensional (3-D) spatial information about metabolism of IMP in regions of the prostate with and without cancer involvement.

After the apparent maximum tolerated dose (MTD) has been established, there will be an expansion of the 3-D imaging cohort to 6 subjects (9 subjects in total at this dose level) to obtain additional information regarding safety at the MTD. If >2 subjects from this cohort of 9 subjects experience a dose-limiting toxicity (DLT), the next lower dose will be defined as the MTD. At the dose level with the highest contrast to noise ratio (dose level less than or equal to the MTD) there will be an expansion of the imaging cohort to include another 15 subjects for a total of 18 subjects who undergo 13C 3-D scanning at this dose, to obtain exploratory information concerning the time course and SNR (signal to noise ratio) of the presence of hyperpolarized [1 13C] pyruvate and its metabolites in regions of cancer and benign prostate tissues. The information provided by these data will be used to develop the MR imaging protocol for future clinical trials that will seek to address the sensitivity and specificity of the technology.

ELIGIBILITY:
INCLUSION CRITERIA:

1. The subject has biopsy-proven prostate cancer and is either undergoing active surveillance ("watchful waiting") or pre primary local treatment for prostate cancer (i.e., prior to either radiation therapy or radical prostatectomy).
2. The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
3. The subject has concordant MRI/1H MRSI findings from a prior MR staging exam performed within 8 weeks of the 13C MRSI exam performed in this study with IMP, or is willing to undergo MRI/1H MRSI in connection with the study exam.
4. Negative test for hepatitis B and hepatitis C.
5. Eastern Cooperative Oncology Group Performance Status of 0 or 1.
6. Laboratory criteria for protocol entry:

   * Absolute neutrophil count (ANC) >/= 1500 cells/microLiters
   * Hemoglobin >/= 9.0 gm/dL
   * Platelets >/= 100,000 cells/microLiters
   * Estimated creatinine clearance >/= 60 mL/min (by the Cockcroft Gault equation)
   * Bilirubin within normal range
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within normal range
7. Willing to use contraception during and for 1 month after completion of the study.

EXCLUSION CRITERIA:

1. The subject has received, or is scheduled to receive, another IMP from 1 month before to 1 month after inclusion in this study.
2. Current or prior androgen deprivation therapy; previous use of a 5-alpha reductase inhibitor is allowed, provided it was discontinued at least 1 month prior to study entry.
3. Poorly controlled hypertension, with blood pressure at study entry >150/90.
4. Contraindication for or inability to tolerate MRI examination.
5. Prostate biopsy within 12 weeks prior to study entry.
6. BMI of less than 18.5 or greater than 32. At the 0.43 ml/kg dose, subject body weight should be less than or equal to 100 kg owing to limitations in the amount of IMP available.
7. Congestive heart failure or New York Heart Association (NYHA) status >2.
8. A past or present medical history of clinically significant electrocardiogram (EKG) abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction (MI) less than 1 year ago with ensuing unstable EKG.
9. Ongoing acute or chronic pulmonary bronchospastic disease, including a history of chronic obstructive pulmonary disease or asthma, with an exacerbation within the past year.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability. | 7 days
  Assessment of the occurrence of clinically significant changes in safety variables from baseline. Safety endpoints include monitoring for the occurrence of treatment-emergent AEs. Monitoring will occur to evaluate for dose-limiting toxicity.
  Dose-Limiting Toxicity (DLT) is defined as any toxicity greater than or equal to grade 2, 3 or 4, attributable to the imaging agent and occurring within 7 days after administration. The maximum tolerated dose will be the dose level at which <33% DLT occurs.

SECONDARY OUTCOMES:
to determine the time course and imaging window that provides the best signal-to-noise ratio (SNR) of the presence of hyperpolarized pyruvate (13C).
  The optimum 13C imaging window for maximizing lactate SNR will be determined as the period of time after injection in which hyperpolarized lactate reaches a maximal plateau in the prostate. This plateau results from opposing processes of lactate production from pyruvate and T1 decay (for pre-clinical studies this plateau occurred approximately between 35 and 55 seconds).
To determine the kinetics and prostate metabolism of hyperpolarized pyruvate (13C)
  For the subjects receiving 3-D 13C spectroscopic imaging (the second 3 subjects per dose cohort as well as the expansion cohorts), a fast 13C MRSI sequence will be used to acquire data from the prostate at a time defined by the kinetic studies (approximately 40 seconds after intravenous administration of hyperpolarized pyruvate).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Albers MJ, Bok R, Chen AP, Cunningham CH, Zierhut ML, Zhang VY, Kohler SJ, Tropp J, Hurd RE, Yen YF, Nelson SJ, Vigneron DB, Kurhanewicz J. Hyperpolarized 13C lactate, pyruvate, and alanine: noninvasive biomarkers for prostate cancer detection and grading. Cancer Res. 2008 Oct 15;68(20):8607-15. doi: 10.1158/0008-5472.CAN-08-0749. PMID 18922937
- [Background] Ardenkjaer-Larsen JH, Fridlund B, Gram A, Hansson G, Hansson L, Lerche MH, Servin R, Thaning M, Golman K. Increase in signal-to-noise ratio of > 10,000 times in liquid-state NMR. Proc Natl Acad Sci U S A. 2003 Sep 2;100(18):10158-63. doi: 10.1073/pnas.1733835100. Epub 2003 Aug 20. PMID 12930897
- [Background] Hricak H, Choyke PL, Eberhardt SC, Leibel SA, Scardino PT. Imaging prostate cancer: a multidisciplinary perspective. Radiology. 2007 Apr;243(1):28-53. doi: 10.1148/radiol.2431030580. PMID 17392247
- [Background] Swanson MG, Zektzer AS, Tabatabai ZL, Simko J, Jarso S, Keshari KR, Schmitt L, Carroll PR, Shinohara K, Vigneron DB, Kurhanewicz J. Quantitative analysis of prostate metabolites using 1H HR-MAS spectroscopy. Magn Reson Med. 2006 Jun;55(6):1257-64. doi: 10.1002/mrm.20909. PMID 16685733
- [Background] Tessem MB, Swanson MG, Keshari KR, Albers MJ, Joun D, Tabatabai ZL, Simko JP, Shinohara K, Nelson SJ, Vigneron DB, Gribbestad IS, Kurhanewicz J. Evaluation of lactate and alanine as metabolic biomarkers of prostate cancer using 1H HR-MAS spectroscopy of biopsy tissues. Magn Reson Med. 2008 Sep;60(3):510-6. doi: 10.1002/mrm.21694. PMID 18727052